CLINICAL TRIAL: NCT06931535
Title: Remote Ischemic Conditioning for Acute Moderate Posterior Ischemic Stroke (RICAMIS2): a Prospective, Random, Open Label, Blinded End Point, Multi-center Study
Brief Title: Remote Ischemic Conditioning for Acute Moderate Posterior Ischemic Stroke
Acronym: RICAMIS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2024) 345
Record Dates: First submitted 2025-04-06; First posted 2025-04-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke
Keywords: posterior circulation stroke; remote ischemic conditioning
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): standard stroke care
- RIC group (Experimental): remote ischemic conditioning, twice a day, for 10 days.
  Interventions: Device: remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — The cuff of the remote ischemic conditioning device was placed on both upper arms (at the same position as blood pressure measurement) and inflated to 200 mmHg. The treatment protocol consisted of 5 cycles of 5-minute inflation followed by 5-minute deflation, performed twice daily. The treatment duration was 8-12 consecutive days.
  Arms: RIC group

SUMMARY:
A substantial body of basic and clinical research has demonstrated the protective effects of remote ischemic conditioning (RIC) in ischemic stroke. While these clinical studies support the safety of RIC, the neuroprotective benefits of RIC in acute ischemic stroke (AIS) patients lack robust evidence due to small sample sizes, heterogeneous RIC protocols, and variability in the severity of neurological deficits among study populations. Our recent multicenter randomized clinical trial, the RICAMIS study, investigated the efficacy of RIC in patients with acute moderate ischemic stroke. The results showed that RIC administered within 48 hours of onset significantly improved 90-day neurological outcomes in patients with moderate stroke severity. It is well established that anterior circulation stroke (ACS) and posterior circulation stroke (PCS) differ in multiple aspects, including anatomical structure, collateral circulation, blood supply, clinical manifestations, prognosis, ischemic tolerance time, and treatment response. For instance, compared to the anterior circulation, the posterior circulation has poorer collateral circulation, a higher proportion of stroke etiologies attributed to atherosclerosis, and longer ischemic tolerance time. Consequently, intravenous thrombolysis and endovascular therapy may offer a more extended therapeutic time window for PCS patients. A prespecified subgroup analysis of the RICAMIS study revealed that patients with PCS derived greater benefit from RIC than those with ACS. However, this finding requires further validation through prospective studies, as prior research has never specifically examined the efficacy of RIC in PCS patients.

Based on the above discussion, this study aims to investigate the efficacy and safety of RIC in patients with acute moderate PCS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Time from onset to treatment: ≤48 hours;
* Posterior circulation ischemic stroke confirmed by CT or MRI, including patients who have received intravenous thrombolysis or endovascular therapy;
* NIHSS score at randomization: 6-16, with an item 1a (level of consciousness) score of 0-1;
* First-ever stroke or prior stroke without significant residual disability (modified Rankin Scale score ≤1);
* Signed informed consent.

Exclusion Criteria:

* intracerebral hemorrhage or subarachnoid hemorrhage；
* Uncontrolled severe hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg despite antihypertensive therapy)；
* Subclavian artery stenosis ≥ 50% or subclavian steal syndrome;
* Intracranial tumor, arteriovenous malformation or aneurysm;
* Severe abnormalities in coagulation;
* Any contraindication for remote ischemic adaptation: the upper limb has serious soft tissue injury, fracture or vascular injury, distal upper limb perivascular lesions, etc.;
* Participating in other clinical trials within 3 months;
* Comorbidity with any serious diseases and life expectancy is less than half a year;
* Patients not suitable for this clinical studies considered by researcher;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
proportion of excellent outcome | 90±7 days
  Excellent outcome is defined as modified Rankin Scale (mRS) score of 0-1. mRS ranges from 0-6, higher scores mean a worse outcome

SECONDARY OUTCOMES:
proportion of favorable outcome | 90±7 days
  Favorable outcome is defined as modified Rankin Scale (mRS) score of 0-2. mRS ranges from 0-6, higher scores mean a worse outcome
Distribution of modified Rankin Scale (mRS) | 90±7 days
  mRS scores range from 0 to 6. mRS ranges from 0-6, higher scores mean a worse outcome.
change in National Institute of Health stroke scale (NIHSS) | 24±6 hours
  NIHSS scores range 0-42, with higher scores indicating greater stroke severity
change in National Institute of Health stroke scale (NIHSS) | 10±2 days
  NIHSS scores range 0-42, with higher scores indicating greater stroke severity
The incidence of stroke-associated pneumonia (SAP) | 10±2 days or during hospitalization, whichever is earlier.
  SAP is defined according to the recommendation from the pneumonia in stroke consensus group (Stroke. 2015; 46:2335-40.)
occurrence rate of the composite events of nonfatal stroke, nonfatal myocardial infarction, and other cardiovascular events | 90±7 days
death due to all causes | 90±7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China